CLINICAL TRIAL: NCT01915082
Title: A Prospective, Randomized, Placebo-controlled Trial of Pre-transplant and Prompt Post-transplant Treatment With Azithromycin to Improve Early Allograft Function and Outcome After Lung Transplantation
Brief Title: Peri-operative Azithromycin to Improve Early Allograft Function and Outcome After Lung Transplantation
Acronym: AZI003
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZI003; 2012-003331-32 (EudraCT Number)
Record Dates: First submitted 2013-07-04; First posted 2013-08-02 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2013-09

CONDITIONS: Disorder Related to Lung Transplantation
Keywords: Lung Function; Allograft Outcome
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin (Experimental): A first dose of azithromycin (25 mL po syrup = 1000 mg) will be given during preparation for subsequent lung transplantation (Day 0).
  After lung transplantation, 'add on' treatment of azithromycin (6.25 mL = 250 mg) syrup will be given via (naso)gastric tube or per os every other day (days 1,3,5,7,9,11,13,15,17,19,21,23,25,27,29 and 31).
  Interventions: Drug: Azithromycin
- Ora-Plus (Placebo Comparator): A first dose of placebo (25 mL po syrup) will be given during preparation for subsequent lung transplantation (Day 0).
  After lung transplantation, 'add on' treatment of placebo (6.25 mL) syrup will be given via (naso)gastric tube or per os every other day (days 1,3,5,7,9,11,13,15,17,19,21,23,25,27,29 and 31).
  Interventions: Drug: Ora-Plus

INTERVENTIONS:
Drug: Azithromycin — Zithromax® oral suspension 200 mg/ 5 mL (Pfizer, UK):
  Zithromax® 1000 mg syrup per os once at recipient intake for lung transplantation (day 0); followed by Zithromax® 250 mg syrup via (naso)gastric tube or per os every other day until one month after lung transplantation (days 1,3,5,7,9,11,13,15, 17,19,21,23,25,27,29 and 31).
  Other Names: Zithromax®
  Arms: Azithromycin
Drug: Ora-Plus — Ora-Plus® oral suspension (Paddock Laboratories, 3940 Quebec Avenue N, Minneapolis, MN 55427, USA; NDC-number: 0574-0303-16):
  Ora-Plus® 25mL syrup per os once at recipient intake for lung transplantation (day 0); followed by Ora-Plus® 6.25 mL syrup via (naso)gastric tube or per os every other day until one month after lung transplantation (days 1,3,5,7,9,11,13,15, 17,19,21,23,25,27,29 and 31).
  Other Names: Ora-Plus®
  Arms: Ora-Plus

SUMMARY:
This study investigates possible beneficial effects of peri-operative treatment (i.e. pre-transplant initiation and prompt post-transplant continuation) with azithromycin in lung transplantation. Our hypothesis is that this therapy will improve early allograft function and outcome following human lung transplantation.

DETAILED DESCRIPTION:
After a lung transplant recipient is put on the waiting list for subsequent lung transplantation, informed consent will be sought for the current study. If signed informed is obtained, the patient will be enrolled upon admission for transplantation at which moment he/she will be randomised to placebo or azithromycin according to a blinded randomisation-list. In accordance with his/her attributed study-number, each included patient will be assigned to a pre-numbered bottle containing the study-drug, which was pre-filled and blinded for its content and are delivered in advance to the ward by the University Leuven Hospital Pharmacy. From this bottle, a first loading dose of placebo (25 mL po syrup) or azithromycin (25 mL po syrup = 1000 mg) will be given by the nurse during preparation for subsequent lung transplantation (Day 0). After lung transplantation, 'add on' treatment of placebo (6.25 mL) or azithromycin (6.25 mL = 250 mg) syrup will be given via (naso)gastric tube or per os every other day (days 1,3,5,7,9,11,13,15,17,19,21,23,25,27,29 and 31) by the nurses taking care of the patient in the early post-transplant period. In case of any serious suspected drug-interactions (however very unlikely) or adverse attributable to the study drug, the study will be promptly stopped in this patient. Serious adverse events will be monitored by the treating lung transplant physicians (blinded for the study-drug) and are defined as allergic reactions including skin reactions (rash, urticaria or Stevens-Johnson syndrome), angioneurotic edema and anaphylaxis, cardiac arrhythmias (ventricular tachycardia or torsades de pointes), neurologic disorders (convulsions). Routine immunosuppressive, prophylactic and necessary antimicrobial treatment according to standardized protocol is given to all patients, independent of study drug. After transplantation, routine follow-up (e.g. biochemical and microbiological blood analyses, chest radiography, pulmonary function testing and bronchoscopic evaluation with broncho-alveolar lavage and/or trans- or endobronchial biopsies will be performed as they are currently routinely being performed as part of the standard, prospective follow-up after lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adult (age at least 18 years old at moment of transplantation)
* Single lung transplantation, sequential single (double) lung transplantation or heart-lung transplantation

Exclusion Criteria:

* Known previous allergy for azithromycin (including skin reactions such as rash, urticaria or Stevens- Johnson syndrome, angioneurotic oedema and anaphylaxis)
* Retransplantation or multi-organ (other than heart-lung) transplantation
* Inclusion in Transmedics® Organ Care System (OCS™ LUNG) study (OCS-LUN-03-2010)(S53795).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mean forced expiratory volume at one second (FEV1, %pred) | at 3 months after lung transplantation
  Mean FEV1 (%pred) during the first 3 months after lung transplantation (measured at discharge; thereafter twice weekly until 8 weeks post-transplant and weekly from 8 to 12 weeks post-transplant; i.e. total estimated number of 14 spirometries per patient)

SECONDARY OUTCOMES:
Length of intubation | at 1 month after lung transplantation
Length of Intensive Care Unit (ICU) stay | at 3 months after lung transplantation
Length of hospital stay | at 3 months after lung transplantation
Partial Pressure of Oxygen in Arterial Blood over fraction of inspired oxygen fraction - ratio (PaO2/FiO2) | at 0, 24, 48 and 72 hours after lung transplantation
Primary graft dysfunction (PGD) prevalence and score | at 0, 24, 48 and 72 hours after lung transplantation
6-minute walking distance | at 1 month after lung transplantation
Acute rejection (grade A; grade B) prevalence/severity | at 1, 3 and 6 months after lung transplantation
Broncho-alveolar lavage neutrophilia and cytokine/protein profile | at day 1 and at 1, 3 and 6 months after lung transplantation
Airway colonization | at day 1 and 1, 3 and 6 months after lung transplantation
  Presence (i.e. growth) of Pseudomonas species or Aspergillus species in routine cultures of broncho-alveolar lavage fluid at day 1 and 1, 3 and 6 months after lung transplantation.
Plasma C-reactive protein levels | at day 1, 3, 5, 7, 14 and 1, 3 and 6 months after lung transplantation
Mortality | at 1, 3 and 6 months after lung transplantation
Ventilator-free days | at 6 months after transplantation
  days alive and free from mechanical ventilation
Mean forced expiratory volume at one second (FEV1, %pred) | at 6 months after lung transplantation
  Mean FEV1 (%pred) during the first 6 months after lung transplantation

OTHER OUTCOMES:
Chronic lung allograft dysfunction | at 1 and 2 years after lung transplantation
Intra-operative respiratory and hemodynamic parameters | at day 1 after lung transplantation
  Intra-operative respiratory parameters (vent. mode (PCV/VCV), Pinsp (PCV), Tidal Volume (VCV/PCV), Ppeak (VCV), Pplat (VCV), Pmean (VCV), PEEP, I:E ratio, One Lung Ventilation (Y/N), Bilateral Lung Ventilation, FiO2, PaO2, PaCO2, End-Tidal CO2, MVSO2) and hemodynamic parameters (PAP (S/D/Mean), BP (S/D/Mean), CO, Heart Rate, CVD) and use of Cardio Pulmonary Bypass or Extra Corporeal Membrane Oxygenation at T0 (after induction) and after 1, 2, 3, 4, 5, 6, 7, 8, etc. hours during transplantation and at the end of operation.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Vos, MD, PhD, Principal Investigator — UZ and KULeuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Van Herck A, Frick AE, Schaevers V, Vranckx A, Verbeken EK, Vanaudenaerde BM, Sacreas A, Heigl T, Neyrinck AP, Van Raemdonck D, Dupont LJ, Yserbyt J, Verleden SE, Verleden GM, Vos R. Azithromycin and early allograft function after lung transplantation: A randomized, controlled trial. J Heart Lung Transplant. 2019 Mar;38(3):252-259. doi: 10.1016/j.healun.2018.12.006. Epub 2018 Dec 14. PMID 30686699